CLINICAL TRIAL: NCT01181830
Title: Effect of Magnesium Administration in Subjects With Family History of Diabetes or Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Cristiano Fava, MD, PhD, Universita di Verona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF_Mg_fam_MetS
Record Dates: First submitted 2010-08-12; First posted 2010-08-13 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Family History of Metabolic Syndrome; Family History of Diabetes
Keywords: magnesium; metabolic syndrome; diabetes; family history
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus | interventions — Pyrrolidonecarboxylic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- magnesium pidolate (Active Comparator): administration of 8.1 mmol bid of magnesium pidolate for 8 weeks
  Interventions: Drug: magnesium pidolate
- placebo (Placebo Comparator): administration of 8.1 mmol bid of placebo for 8 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: magnesium pidolate — administration of 8.1 mmol bid of magnesium pidolate
  Arms: magnesium pidolate
Drug: placebo — administration of 8.1 mmol bid of placebo
  Arms: placebo

SUMMARY:
Magnesium is the second most abundant ion in human cells and plays fundamental roles in several enzymatic reactions: it is involved in ATP production, in the phosphorylation of proteins, in glucose metabolism and in the contraction of cytoskeleton.

Several epidemiological studies demonstrated that low dietary magnesium intake is inversely associated with diabetes mellitus, hypertension and metabolic syndrome.

Magnesium could be related to important haemodynamic and metabolic anomalies: at vascular level it acts as an antagonist of calcium, especially in vascular smooth muscle cells, thus its deficit could enhance vascular contraction; with regard to glucose metabolism, magnesium is involved in the physiopathological mechanism of insulin resistance, through a reduction in cellular uptake of glucose. This condition and the subsequent compensatory hyperinsulinemia can ultimately lead to increased synthesis of proinflammatory cytokines and to endothelial dysfunction. Thus, magnesium depletion and subsequent alterations can increase the risk of developing vascular disease such as atherosclerosis and has been associated with cardiovascular events.

Several clinical trials have explored the possible beneficial effect of magnesium supplementation on blood pressure, plasma lipids and insulin resistance but the results are often contradictory. One of the possibilities for these unclear results could be that in some of them the interventions started too late when haemodynamic and metabolic changes are more difficult to revert.

The investigators hypothesis is that magnesium supplementation in a population at increased genetic risk of developing metabolic syndrome but without it could improve blood pressure and the other metabolic syndrome related components.

Thus, the aim of the present study is to evaluate the effect of oral supplementation of magnesium (16.2 mmol/day of magnesium pidolate) on metabolic syndrome's components in a sample of 15 subjects who are at increased risk of developing metabolic syndrome since have a positive familiar history of type II diabetes mellitus and/or metabolic syndrome(AHA/NHLBI criteria).

ELIGIBILITY:
Inclusion Criteria:

* positive family history of type II diabetes mellitus and/or metabolic syndrome(AHA/NHLBI criteria).

Exclusion Criteria:

* any therapy related to metabolic syndrome (that is antihypertensive, anti diabetic, antilipemic drugs);
* age < 18 years or >50 years;
* previously diagnosed hypertension or immediate need for antihypertensive therapy (BP≥160/100);
* diabetes mellitus (ADA criteria);
* obesity (BMI>30Kg/m2);
* Continuative use of NSAIDs, magnesium or vitamin supplements;
* Hypermagnesaemia;
* Previous cardio- or cerebrovascular events;
* chronic kidney or liver or inflammatory or neoplastic disease;
* gastrointestinal dysfunction with hypomotility;
* active smoke (>5 cigarettes per day);
* Impossibility to give informed consent.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 8 weeks
  Blood pressure measured in the lying and standing position (average of three measurements);

SECONDARY OUTCOMES:
other features of metabolic syndrome | 8 weeks
  especially plasma lipids and HOMA index
endothelial function | 8 weeks
  endothelial function as measured non-invasively by ultrasound using the "Flow Mediated Dilatation" (FMD) technique
arterial stiffness | 8 weeks
  systemic and local arterial stiffness measured by digital photoplethysmography and by carotid ultrasound
Inflammation | 8 weeks
  Markers of inflammation such as C reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Delva, MD, Principal Investigator — Universita of Verona; Cristiano Fava, MD, PhD, Principal Investigator — Universita of Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata - Division of Internal Medicine C, Verona, VR, Italy

REFERENCES:
- [Derived] Cosaro E, Bonafini S, Montagnana M, Danese E, Trettene MS, Minuz P, Delva P, Fava C. Effects of magnesium supplements on blood pressure, endothelial function and metabolic parameters in healthy young men with a family history of metabolic syndrome. Nutr Metab Cardiovasc Dis. 2014 Nov;24(11):1213-20. doi: 10.1016/j.numecd.2014.05.010. Epub 2014 May 28. PMID 24984823